CLINICAL TRIAL: NCT06205355
Title: Comparison of Goal-directed Analgesia Using ANI (Analgesia/Nociception Index) and Standard Analgesia During General Anesthesia in Patients Undergoing Orthognathic Surgery on Postoperative Quality of Recovery: a Prospective Randomized Controlled Trial
Brief Title: Analgesia Nociception Index in Orthognathic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-2310-152-1481
Record Dates: First submitted 2023-12-13; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- goal-directed analgesia using ANI monitoring (Experimental)
  Interventions: Device: Analgesia/Nociception Index (ANI) monitoring
- Standard monitoring (Active Comparator)
  Interventions: Device: Standard monitoring

INTERVENTIONS:
Device: Analgesia/Nociception Index (ANI) monitoring — intraoperative analgesia was provided by infusion of remifentanil via target controlled infusion mode, which was controlled according to ANI monitor.
  Arms: goal-directed analgesia using ANI monitoring
Device: Standard monitoring — intraoperative analgesia was provided by infusion of remifentanil via target controlled infusion mode, which was controlled according to the clinician's decision
  Arms: Standard monitoring

SUMMARY:
This study aims to determine whether goal-directed analgesia using ANI(Analgesia/Nociception Index) can improve the quality of postoperative recovery in patients undergoing maxillofacial surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 or older undergoing maxillary, mandibular, or bimaxillary surgery under general anesthesia.
* adult patients who can provide written informed consent to participate in the study, understand the procedures of this study, and be able to complete patient-reported questionnaires adequately.
* adult patients who Have made an informed decision to participate in this study and have given written consent.

Exclusion Criteria:

* Patients with ASA physical status 4-5
* Emergency surgery
* Patients with chronic pain and related pain medications
* Patients with hypersensitivity to general anesthesia drugs and pain medications
* Patients with arrhythmia
* Pregnant women
* Others deemed unsuitable by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative QoR-15K score | 24 hours after the end of surgery
  Korean-translated QoR-15K (15-item Quality of Recovery (QoR-15) scale, minimum 0, maximum 150, higher scores mean a better outcome ) scores assessed by participants blinded to arm assignment 24 hours after surgery.

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours after the end of surgery
  Postoperative satisfaction as assessed by study participants blinded to group assignment, recorded on an NRS scale from a low of 0 to a high of 10.
intraoperative opioid consumption | during surgery
  total dose of remifentanil consumption during surgery
intraoperative non-opioid consumption | during surgery
  total dose of non-opioid consumption during surgery
intraoperative use of vasoactive drugs | during surgery
  total dose of vasoactive drugs during surgery
The time-weighted average of the segments of the total anesthesia time where the ANI value did not remain above 50 and below 70. | during surgery
Percentage of time with a deviation of more than ±20% from the mean blood pressure measured on the ward as a percentage of total anesthesia time | during surgery
estimated blood loss | during surgery
total fluid administration during surgery | during surgery
extubation time | from the end of surgery to endotracheal tube extubation, up to 30 minutes
number of participants with postoperative nausea vomiting | 24 hours after the end of surgery
number of participants with postoperative opioid-related side effects (constipation, pruritis, dizziness, dry mouth, somnolence) | 24 hours after the end of surgery
Total postoperative opioid consumption | 24 hours after the end of surgery
Total postoperative non-opioid consumption | 24 hours after the end of surgery
postoperative pain measured by numerical rating scale (NRS) scale (minimum 0, maximum 10, higher scores mean worse outcome) | 24 hours after the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea